CLINICAL TRIAL: NCT00726050
Title: The Relationship Between Temporal Discrimination and Cortical Excitability in Humans
Brief Title: Brain Activity in Time Discrimination and Sensory Input
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080189; 08-N-0189
Record Dates: First submitted 2008-07-30; First posted 2008-07-31 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-04-29

CONDITIONS: Healthy Volunteers
Keywords: Theta Burst Stimulation; Somatosensory Stimulation; Somatosensory Cortex; Tactile Discrimination; Healthy Volunteer; HV

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will use repetitive transcranial magnetic stimulation, or rTMS (magnetic stimulation to the brain), to examine how the brain distinguishes between two signals that are spaced very closely in time. The ability to tell the difference between sensory signals is important to understanding sensory input. Understanding how this works may help to develop new treatments for sensory deficits.

Healthy volunteers 18 years of age and older may be eligible for this study. Participants undergo the following procedures during three visits to the NIH Clinical Center:

rTMS - all visits (sham rTMS on one visit) :

For TMS, a wire coil is held on the scalp. A brief electrical current passed through the coil creates a magnetic pulse that stimulates the brain. During the stimulation, the subject may be asked to tense certain muscles slightly or perform other simple actions.

Theta burst stimulation (TBS) - all visits (sham TBS on one visit):

Same as TMS, but brief pulses of electrical current are passed through the coil. Subjects undergo intermittent TBS on one visit and continuous TBS on another.

Somatosensory evoked potential (SEP) - all visits:

SEP tests how sensory information travels along the nerves to the spinal cord and brain. A small metal disk electrode placed on an arm delivers a small electrical shock. Electrodes placed on the scalp record how the impulse travels over the nerve pathways to the cerebral cortex of the brain. EEG (see below) records what sensory information the brain is detecting and processing. Paired-pulse SEP is done before and after TBS.

Temporal discrimination threshold - all visits:

This test investigates the brain's ability to discriminate sensory information. Electrodes are placed on the subject's wrist. Two electrical pulses are delivered to the nerve at the wrist at different spaced intervals to determine when the subject feels the two pulses are fused into one. This test is done before and after TBS.

Electroencephalography (EEG) - all visits:

This test records brain waves (electrical activity of the brain). Electrodes are placed on the scalp with an electrode cap. The spaces between the electrodes and the scalp are filled with a gel that conducts electrical activity.

DETAILED DESCRIPTION:
Objective:

The ability to discriminate successive signals separated by time intervals in the millisecond-range is an important element in analyzing the temporal characteristics of sensory input. When two identical stimuli are presented with a sufficient time interval between them, they are readily perceived as being two separate events. As they are presented progressively closer together, there comes a point when the two separate stimuli are perceived as one. However, the neural mechanism of temporal discrimination is unclear. Therefore, our major objective is to analyze, in detail, the effect of cortical excitability and inhibition on temporal sensory discrimination in healthy subjects.

Study Population:

We intend to study 25 adult healthy volunteers.

Design:

Assuming the cortical circuit in the somatosensory area plays an important role in temporal discrimination, we plan to investigate the relationship between cortical excitability and the ability of temporal discrimination. We hypothesize that the extent of cortical excitability affects the ability to discriminate. Cortical excitability will be modulated by using repetitive transcranial magnetic stimulation (rTMS). Comparison of cortical excitability changes will be determined before and after rTMS in the primary somatosensory cortex (SI). The change in cortical information processing in SI will be studied using multi-channel electroencephalography (EEG) recording of paired-pulse somatosensory evoked potentials (SEPs) delivered at rest. Activity assessment in the cortical circuit will be measured by the recovery curve of the amplitude of paired-pulse SEPs.

Outcome Measures:

The primary outcome measure will be the change in amplitude of the paired-pulse SEP component (P27) in 5-ms interstimulus interval condition for three types of rTMS. The secondary outcome will be the amplitude of paired-pulse SEP components during other interstimulus interval conditions (10 to 200 ms).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 years and older
* Absence of dystonia or other neurological conditions

EXCLUSION CRITERIA:

* Concurrent medical, surgical, neurologic or psychiatric condition
* History of neurological disorders
* History of seizure disorder
* Pregnant women
* Presence of pacemaker, implanted medical pump, metal plate or metal object in skull or eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-07-28; Study Completion 2010-04-29

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aglioti SM, Fiorio M, Forster B, Tinazzi M. Temporal discrimination of cross-modal and unimodal stimuli in generalized dystonia. Neurology. 2003 Mar 11;60(5):782-5. doi: 10.1212/01.wnl.0000046528.24693.5b. PMID 12629233
- [Background] Akatsuka K, Wasaka T, Nakata H, Inui K, Hoshiyama M, Kakigi R. Mismatch responses related to temporal discrimination of somatosensory stimulation. Clin Neurophysiol. 2005 Aug;116(8):1930-7. doi: 10.1016/j.clinph.2005.04.021. PMID 15982927
- [Background] Angel A. Cortical responses to paired stimuli applied peripherally & at sites along the somato-sensory pathway. J Physiol. 1967 Jul;191(2):427-48. doi: 10.1113/jphysiol.1967.sp008260. PMID 6050113